CLINICAL TRIAL: NCT04901585
Title: Enterotomy Closure After Minimally Invasive Distal Gastrectomy With Intracorporeal Anastomosis.
Brief Title: Enterotomy Closure and Minimally Invasive Gastrectomy
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Milone, Professor, Federico II University
Other Study IDs: intragastrectomy
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Gastric Cancer
Keywords: intracorporeal gastrectomy; enterotomy closure
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Totally intracorporeal distal gastrectomy: All patients who underwent minimally invasive distal gastrectomy with intracorporeal anastomosis for gastric cancer
  Interventions: Procedure: Totally intracorporeal distal gastrectomy

INTERVENTIONS:
Procedure: Totally intracorporeal distal gastrectomy — Minimally invasive distal gastrectomy with intracorporeal anastomosis and handsewn enterotomy closure

SUMMARY:
All consecutive patients from January 2009 to december 2019 who underwent minimally invasive partial gastrectomy for gastric cancer at thirteen high volume institutions will be retrospective analysed to assess the better way to fashion a handsewn intracorporeal enterotomy closure after a stapled anastomosis.

DETAILED DESCRIPTION:
Different ways to fashion intracorporeal anstomoses will be investigated: robotic vs laparoscopic approach; laparoscopic HD vs 3D vs 4K technologies; single layer vs double layer enterotomy closure. Additionally double layer enterotomies will be analysed layer by layer, comparing running vs interrupted suture, presence vs absence of deep corner suture and type of suture thread (barbed, braided, non braided suture)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* laparoscopic or robotic partial gastrectomy for gastric cancer
* Roux en Y or Billroth II reconstruction

Exclusion Criteria:

* Age < 18 years
* open gastrectomy
* total gastrectomy
* Billroth I reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent laparoscopic or robotic partial gastrectomy for gastric cancer with Roux en Y or Billroth II reconstruction
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 1 month
  The better way to fashion enterotomy closure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy